CLINICAL TRIAL: NCT05236660
Title: Cost-utility of an Integrated Personalised Assistive Devices Approach to Reduce Foot Ulcer Recurrence in Diabetes (DIASSIST): a Multicentre Randomised Controlled Trial
Brief Title: Personalised Assistive Devices Approach for Diabetic Foot Ulcer Prevention
Acronym: DIASSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Sicco Bus, PhD, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL78943.018.21
Record Dates: First submitted 2022-01-17; First posted 2022-02-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetes; foot ulcer; prevention; cost-utility
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal care (Experimental): Multimodal personalised treatment
  Interventions: Device: Custom-made shoes: pressure-optimized; Device: Custom-made indoor shoes: pressure optimized; Device: Foot temperature monitoring; Behavioral: Education
- Usual care (No Intervention): Usual care as offered to high-risk patients as offered in the Netherlands

INTERVENTIONS:
Device: Custom-made shoes: pressure-optimized — Pressure-optimized custom-made shoes: evaluated and optimized using in-shoe pressure analysis, and re-evaluated after 6 months.
  Arms: Multimodal care
Device: Custom-made indoor shoes: pressure optimized — Pressure-optimized custom-made indoor shoes: evaluated and optimized using in-shoe pressure analysis, and re-evaluated after 6 months. Specifically designed for indoor use.
  Arms: Multimodal care
Device: Foot temperature monitoring — Personalised at-home daily foot temperature monitoring at high-risk regions.
  Arms: Multimodal care
Behavioral: Education — Personalised patient education consisting of quantitative feedback on in-shoe pressures, temperature measurements and footwear use and, in addition, motivational interviewing where indicated and needed to improve device use.
  Arms: Multimodal care

SUMMARY:
Preventing foot ulcers in people with diabetes can reduce costs and increase quality of life. Despite availability of various interventions to prevent foot ulcers, recurrence rates remain high. We hypothesise that a multimodal approach incorporating a variety of orthotic interventions that matches an individual person's need can reduce ulcer recurrence with beneficial cost-effectiveness and cost-utility.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2
* Age 18 years or above
* Loss of protective sensation based on the presence of peripheral neuropathy
* A healed plantar foot ulcer or foot amputation in the preceding 4 years until two weeks before study inclusion
* In possession of custom-made orthopaedic shoes, defined as "Orthopaedic shoes type A" or "Orthopaedic shoes type B" , or Orthopaedic Provision in Regular Footwear (OVAC), according to the Dutch healthcare system
* Ability to provide informed consent

Exclusion Criteria:

* Foot ulcer or open amputation site(s)
* Active Charcot's neuroarthropathy
* Foot infection, based on criteria of the PEDIS classification
* Amputation proximal to the metatarsal bones in both feet
* Healed ulcer on the apex of digitus 2-5 as the only ulcer location in the past 4 years, as surgical intervention (flexor tenotomy) is a more likely and guideline-recommended treatment for such patients, rather than the multimodal care under investigation
* Severe illness that would make 12-months survival unlikely, based on the clinical judgment by the physician
* Concomitant severe physical or mental conditions that limit the ability to follow instructions for the study, based on clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Cost-utility (as the primary economic outcome) | 12 months (full study period)
  defined as the ratio between costs related to foot care and quality-adjusted life years, based on the health utilities associated with the scoring profiles on the EQ-5D-5L with Dutch reference scores
Adherence to wearing custom-made footwear (as the primary patient-related outcome) | 12 months (full study period)
  defined as the percentage of steps taken in prescribed footwear, calculated by combining physical activity and wearing time measurements
Foot ulcer recurrence during the 12-months follow-up (as the primary clinical outcome) | 12 months (full study period)
  defined as "a break of the skin of the foot that involves as a minimum the epidermis and part of the dermis, in a person who has a history of foot ulceration, irrespective of location and time since the previous foot ulcer", with the first ulcer in the study period recorded as primary outcome and percentage participants with ulcer recurrence on group level as primary outcome

SECONDARY OUTCOMES:
Cost-effectiveness | 12 months (full study period)
  defined as the ratio between costs related to foot care and foot ulcer recurrence on any location of the foot
Plantar foot ulcer recurrence | 12 months (full study period)
  following the definition of foot ulcer recurrence (outcome 3), but then limited to the plantar side of the foot
Foot ulcer recurrence at three predefined high-risk locations | 12 months (full study period)
  following the definition of foot ulcer recurrence (outcome 3), but then limited to a maximum 3 high risk locations per participant, specified at the start of the study, based on barefoot pressures, ulcer history, pre-ulcerative lesions or signs of abundant callus
Costs related to foot care (from a societal and medical perspective) | 12 months (full study period)
  Costs will be calculated for each participant as the product sum of resource volume data and their respective unit costs. Resource volume data will be obtained from the completed study specific versions of the institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ) and iMTA Productivity Cost Questionnaire (iPCQ), as these contain the volume data on healthcare resource utilization, out-of-pocket expenses and loss of productivity related to foot care. Foot care includes both care for ulcer prevention (e.g. podiatry appointments, rehabilitation physician consultations) and for ulcer treatment (e.g. multidisciplinary treatment, hospitalization, surgery). Reference prices for unit costs will be based on the most recent Dutch manual for costing in healthcare research available at the time of analysis. All costs will be summed during the entire study period.
Quality-adjusted life years | 12 months (full study period)
  based on the health utilities associated with the scoring profiles on the EQ-5D-5L with Dutch reference scores. This will be monitored during the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sicco Bus, Prof, Principal Investigator — Amsterdam UMC
Locations (5):
- Netherlands (5):
  - Amsterdam UMC, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Reinier de Graaf Gasthuis, Delft
  - Spaarne Gasthuis, Hoofddorp
  - Máxima Medisch Centrum, Veldhoven

IPD SHARING:
Plan to Share IPD: Yes
Data can be made available after an embargo period, to allow the research team to write all prespecified publications. The embargo period is required, as publications may often follow once the project has already ended. The embargo period will be a maximum 2 years, to allow the research sufficient time to finish the publications as specified in the protocol. If publications are available earlier, the embargo will end earlier.
  Conditions for reuse will apply, but have yet to be finalized.
Supporting Information: Study Protocol
Time Frame: 2 years after study completion and for 15 years
Access Criteria: to be determined

REFERENCES:
- [Derived] Vossen LE, van Netten JJ, Bakker CD, Berendsen HA, Busch-Westbroek TE, Peters EJG, Sabelis LWE, Dijkgraaf MGW, Bus SA. An integrated personalized assistive devices approach to reduce the risk of foot ulcer recurrence in diabetes (DIASSIST): study protocol for a multicenter randomized controlled trial. Trials. 2023 Oct 12;24(1):663. doi: 10.1186/s13063-023-07635-z. PMID 37828618